CLINICAL TRIAL: NCT02069613
Title: Multimodal Approach to Testing the Acute Effects of Mild Traumatic Brain Injury (mTBI)
Status: Completed | Type: Observational
Sponsor: Huntington Medical Research Institutes (Other)
Collaborators: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael G Harrington, Research Scientist, Huntington Medical Research Institutes
Other Study IDs: 27294/1; W81XWH-13-1-0005 (Other Grant/Funding Number: USAMRMC)
Record Dates: First submitted 2014-02-18; First posted 2014-02-24 (Estimated); Last update posted 2017-11-08 (Actual); Status verified 2017-11

CONDITIONS: Concussion, Mild
Keywords: Mild traumatic injury to extremity (for controls); mTBI; concussion; MEG; EEG; Blood; MRI; DTI; biomarkers
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood will be retained for future analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Mild traumatic brain injury (mTBI): Patients admitted to Huntington Memorial Hospital (HMH), Pasadena CA, Emergency Department (ED) diagnosed with mTBI by history (alteration of consciousness, post-traumatic amnesia, loss of consciousness) and normal brain computed tomography (CT).
- Control: Patients admitted to HMH ED for minor extremity trauma (sprains) and no evidence of mTBI

SUMMARY:
The objective of the study is to determine the relative roles for various testing modalities in the diagnosis and prognosis of mild traumatic brain injury.

DETAILED DESCRIPTION:
Subjects will undergo functional brain testing (magnetoencephalography, electroencephalography), anatomical brain imaging (diffusion tensor imaging, susceptibility-weighted imaging), neuropsychological testing (memory, language, processing speed), sleep patterns using actigraphy, and blood testing of candidate biomarkers. Testing will be done at 3 time points post-injury: 1 day, 14 days, and 30 days post-injury. Analysis of these tests collectively will be used to develop diagnostic tools for acute mTBI.

ELIGIBILITY:
Inclusion Criteria:

1. Civilian (non-military) presenting to HMH ED.

Exclusion Criteria:

1. Prior history of diagnosed TBI.
2. Other significant non-head injury/trauma or open wound.
3. Other significant medical co-morbidities, such as heart disease or cancer.
4. Self-reported current use or substances contributing to ED visit (e.g. illicit drugs, medications, alcohol abuse).
5. Currently diagnosed psychological condition (e.g. depression, PTSD).
6. Medications for psychological or neurological disorder.
7. Any implanted metal, such as medical device or braces on teeth.
8. Injury to the back or other injury that will make it difficult for the participant to tolerate tests.
9. Injury to dominant arm that would cause difficulty using computer or responding to stimuli during functional imaging.
10. Pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Study participants (control, mTBI) will be referred by the Huntington Hospital Emergency Department staff. ED staff will determine the eligibility criteria. If consent is achieved, testing will occur at pre-determined times: 1 day, 14 days, and 30 days post-injury.
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2014-03; Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Change in objective measures of brain function (MEG/EEG, blood biomarkers) | Day 1, day 14, and day 30 post-injury
  For MEG/EEG, resting state analyses of brain function will be conducted to include frequency band analyses localizing, for example, delta slow wave activity, and establishing functional connectivity scores at three time points post injury (day 1, day 14, day 30). For blood biomarkers, serum levels in approximately ten biomarkers will be measured to determine amount in each and if changes occur at three time points post-injury.

SECONDARY OUTCOMES:
Change in anatomical measures of brain function (DTI, SWI) | Day 1, day 14, and day 30 post-injury
  Diffusion Tensor-derived measures will be calculated for control and mTBI participants to determine if changes occur at three time points post-injury (day 1, day 14, day 30).

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Harrington, MB, Principal Investigator — Huntington Medical Research Institutes
Locations (3):
- United States (3):
  - Huntington Medical Research Institutes, Pasadena, California
  - HMRI, Pasadena, California
  - Molecular Neurology Program, Pasadena, California

REFERENCES:
- [Background] Hoge CW, McGurk D, Thomas JL, Cox AL, Engel CC, Castro CA. Mild traumatic brain injury in U.S. Soldiers returning from Iraq. N Engl J Med. 2008 Jan 31;358(5):453-63. doi: 10.1056/NEJMoa072972. Epub 2008 Jan 30. PMID 18234750
- [Background] Bigler ED. Neuropsychology and clinical neuroscience of persistent post-concussive syndrome. J Int Neuropsychol Soc. 2008 Jan;14(1):1-22. doi: 10.1017/S135561770808017X. PMID 18078527
- [Background] Lewine JD, Davis JT, Bigler ED, Thoma R, Hill D, Funke M, Sloan JH, Hall S, Orrison WW. Objective documentation of traumatic brain injury subsequent to mild head trauma: multimodal brain imaging with MEG, SPECT, and MRI. J Head Trauma Rehabil. 2007 May-Jun;22(3):141-55. doi: 10.1097/01.HTR.0000271115.29954.27. PMID 17510590
- [Background] Huang MX, Theilmann RJ, Robb A, Angeles A, Nichols S, Drake A, D'Andrea J, Levy M, Holland M, Song T, Ge S, Hwang E, Yoo K, Cui L, Baker DG, Trauner D, Coimbra R, Lee RR. Integrated imaging approach with MEG and DTI to detect mild traumatic brain injury in military and civilian patients. J Neurotrauma. 2009 Aug;26(8):1213-26. doi: 10.1089/neu.2008.0672. PMID 19385722
- [Background] Pelinka LE, Kroepfl A, Schmidhammer R, Krenn M, Buchinger W, Redl H, Raabe A. Glial fibrillary acidic protein in serum after traumatic brain injury and multiple trauma. J Trauma. 2004 Nov;57(5):1006-12. doi: 10.1097/01.ta.0000108998.48026.c3. PMID 15580024
- [Background] Vos PE, Lamers KJ, Hendriks JC, van Haaren M, Beems T, Zimmerman C, van Geel W, de Reus H, Biert J, Verbeek MM. Glial and neuronal proteins in serum predict outcome after severe traumatic brain injury. Neurology. 2004 Apr 27;62(8):1303-10. doi: 10.1212/01.wnl.0000120550.00643.dc. PMID 15111666